CLINICAL TRIAL: NCT07010159
Title: A Phase 2/3 Efficacy and Safety Study of KPL-387 Treatment in Participants With Recurrent Pericarditis
Brief Title: Phase 2/3 Study of KPL-387 in Recurrent Pericarditis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals International, plc (Industry)
Collaborators: Kiniksa Pharmaceuticals, GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KPL-387-C211; 2025-521933-10 (EudraCT Number)
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Pericarditis; Pericarditis Acute; Recurrent Pericarditis
Keywords: Recurrence; Recurrent; Recurrent Pericarditis; KPL-387
MeSH Terms: conditions — Pericarditis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 2 KPL-387 100mg SC q2wk (Experimental): In Phase 2 Treatment Period KPL-387 will be administered by subcutaneous (SC) injection every 2 weeks (q2wk) through Week 22.
  Interventions: Drug: KPL-387
- Phase 2 KPL-387 100mg SC q4wk (Experimental): In Phase 2 Treatment Period, KPL-387 or placebo (alternating every 2 weeks) will be administered by SC injection q2wk through Week 22 to provide active drug administration every 4 weeks (q4wk) while maintaining treatment concealment.
  Interventions: Drug: KPL-387; Drug: Placebo
- Phase 2 KPL-387 300mg SC q2wk (Experimental): In Phase 2 Treatment Period KPL-387 will be administered by SC injection q2wk through Week 22.
  Interventions: Drug: KPL-387
- Phase 2 KPL-387 300mg SC q4wk (Experimental): In Phase 2 Treatment Period, KPL-387 or placebo (alternating every 2 weeks) will be administered by SC injection q2wk through Week 22 to provide active drug administration q4wk while maintaining treatment concealment.
  Interventions: Drug: KPL-387; Drug: Placebo
- Phase 3 KPL-387 SC (Experimental): Run-In (RI) Period: participants receive single-blind KPL-387
  Randomized Withdrawal (RW) Period: eligible participants are randomized (1:1 KPL-387 or placebo) to receive double-blinded KPL-387.
  Interventions: Drug: KPL-387
- Phase 3 Placebo SC (Placebo Comparator): RW Period: eligible participants are randomized (1:1 KPL-387 or placebo) to receive double-blinded placebo.
  Interventions: Drug: Placebo
- Long-Term Extension (Experimental): Participants from Phase 2 and Phase 3 who continue into the Long-Term Extension will receive KPL-387.
  Interventions: Drug: KPL-387

INTERVENTIONS:
Drug: KPL-387 — administered by subcutaneous injection
  Arms: Long-Term Extension; Phase 2 KPL-387 100mg SC q2wk; Phase 2 KPL-387 100mg SC q4wk; Phase 2 KPL-387 300mg SC q2wk; Phase 2 KPL-387 300mg SC q4wk; Phase 3 KPL-387 SC
Drug: Placebo — administered by subcutaneous injection
  Arms: Phase 2 KPL-387 100mg SC q4wk; Phase 2 KPL-387 300mg SC q4wk; Phase 3 Placebo SC

SUMMARY:
This study is being done to demonstrate whether KPL-387 is an effective and safe treatment for recurrent pericarditis.

DETAILED DESCRIPTION:
This clinical trial is comprised of 3 separate study parts: Phase 2, Phase 3, and Long-Term Extension. The primary objective of Phase 2 is to evaluate how well different dose regimens of KPL-387 control the pain and inflammation of pericarditis in a group of participants experiencing an acute episode of recurrent pericarditis. This part of the study will confirm the KPL-387 dose regimen to be further tested in Phase 3 and the Long-Term Extension. The primary objective of Phase 3 is to confirm the efficacy of KPL-387 for the treatment of recurrent pericarditis and reduction in risk of recurrence in an additional group of participants experiencing an acute episode of recurrent pericarditis. Participants who complete Phase 2 or Phase 3 may be eligible to participate in the Long-Term Extension. The primary objective of the Long-Term Extension is to assess the long-term efficacy of KPL-387 while maintaining long-term disease control. All of the study parts also have other objectives to learn about the safety, tolerability, concentration of KPL-387 in blood, and effects of KPL-387 on blood test markers of immune activity in recurrent pericarditis.

ELIGIBILITY:
Key Inclusion Criteria:

* Phase 2 and 3: Has a diagnosis of recurrent pericarditis
* Phase 2 and 3: Has signs and symptoms of recurrent pericarditis despite treatment with standard therapies
* Phase 2 and 3: Weighs at least 40 kg
* Phase 2: Taking NSAIDS and/or colchicine (in any combination)
* Phase 3: Taking NSAIDs and/or colchicine and/or glucocorticoids (in any combination)

Key Exclusion Criteria:

* Phase 2 and 3: Has a diagnosis of pericarditis that is secondary to specific prohibited etiologies.
* Phase 2 and 3: Has received an investigational drug during the 4 weeks before screening or is planning to receive an investigational drug at any time during the study.
* Phase 2 and 3: Has a history of active or untreated, latent tuberculosis (TB) prior to screening.
* Phase 2 and 3: Has a history of immunodeficiency.
* Phase 2 and 3: Has a history of immunosuppression, including positive human immunodeficiency virus (HIV) test results.
* Phase 2 and 3: Has chest x-ray at Screening or within 12 weeks before first study drug administration, with evidence of malignancy, abnormality consistent with prior or active TB infection or active infection.
* Phase 2 and 3: Has a history of malignancy of any organ system within the past 5 years before Screening (other than a successfully treated non metastatic cutaneous squamous cell carcinoma or basal cell carcinoma and/or localized carcinoma in situ of the cervix).
* Phase 2 and 3: Has a known or suspected current active infection or a history of chronic or recurrent infectious disease (> 3 episodes in prior 12 months), including but not limited to, genitourinary infection, chest infection, sinusitis, or skin/soft tissue infection.
* Phase 2 and 3: Has had a serious infection, has been admitted to the hospital for an infection, or has been treated for a documented infection requiring antibiotics for a documented infection within 2 weeks prior to first study drug administration.
* Phase 2 and 3: Has had an organ transplant (except corneal transplant performed more than 3 months prior to first study drug administration).
* Phase 2 and 3: In the Investigator's opinion, has any other medical condition that could adversely affect the subject's participation or interfere with study evaluations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Time to Treatment Response by Week 24 | From Randomization up to Week 24
Phase 3: Time to Pericarditis Recurrence | From first administration of study drug in the RW Period
Long-Term Extension: Annualized rate of Pericarditis Recurrence | Up to 24 Months

SECONDARY OUTCOMES:
Phase 2: Time to CRP Normalization (CRP ≤ 0.5 mg/dL) by Week 24 | From Randomization up to Week 24
Phase 2: Time to Pain Response by Week 24 | From Randomization up to Week 24
Phase 2: Percentage of Days With No or Minimal Pain (Numerical Rating Scale (NRS) ≤ 2) While on KPL-387 Treatment Over Time by Week 24 | From Randomization up to Week 24
Phase 2: Proportion of Participants With Normalization of CRP (CRP ≤ 0.5 mg/dL) Over Time by Week 24 | From Randomization up to Week 24
Phase 2: Time to resolution of pericarditis manifestations (i.e. echocardiogram [ECHO] abnormalities, electrocardiogram [ECG] abnormalities, and pericardial rub), when present at Baseline, by Week 16. | From Randomization up to Week 16
Phase 2: Change from Baseline in SF-36v2® Physical Component Summary score through Week 24. | From Randomization up to Week 24
Phase 2: Change from Baseline in SF-36v2® Mental Component Summary score through Week 24. | From Randomization to Week 24
Phase 2: Proportion of participants with Protocol-Defined Pericarditis Recurrence by Week 24. | From Randomization to Week 24
Phase 2: Change from Baseline in CRP through Week 24. | From Randomization up to Week 24
Phase 2: Change from Baseline in pericarditis pain NRS score through Week 24. | From Randomization up to Week 24
Phase 2: Change from RI Baseline in SF-36v2® Mental Component Summary score through the end of the RI Period | From Baseline up to the end of the RI Period
Phase 3: Time to Treatment Response by the end of the RI Period | From Baseline up to end of the RI Period
Phase 3: Time to Clinical Response by the end of the RI Period | From Baseline up to end of the RI Period
Phase 3: Time to Pain Response by end of the RI Period | From Baseline up to end of the RI Period
Phase 3: Time to CRP normalization by the end of the RI Period | From Baseline up to end of the RI Period
Phase 3: Change from RI Baseline in SF-36v2® Physical Component Summary score through the end of the RI Period. | From Baseline up to end of the RI Period
Phase 3: Time to resolution of pericarditis manifestations (i.e., ECHO abnormalities, ECG abnormalities, and pericardial rub), when present at RI Baseline, by the end of the RI period. | From Baseline up to end of the RI Period
Phase 3: Change from RI Baseline in daily pericarditis pain NRS score through the end of the RI Period. | From Baseline up to end of the RI Period
Phase 3: Change from RI Baseline in CRP through the end of the RI Period. | From Baseline up to end of the RI Period
Phase 3: Proportion of participants who maintained Clinical Response at RW Week 16. | From Randomization up to RW Week 16
Phase 3: Percentage of days with no or minimal pericarditis pain through RW Week 16. | From Randomization up to RW Week 16
Phase 3: Change from RW Baseline in SF-36v2® Physical Component Summary score at RW Week 16. | From Randomization up to RW Week 16
Phase 3: Change from RW Baseline in SF-36v2® Mental Component Summary score at RW Week 16 | From Randomization up to RW Week 16
Phase 3: Change from RW Baseline in pain NRS score during the RW Period. | From Randomization through the end of the RW Period
Phase 3: Change from RW Baseline in CRP during the RW Period | From Randomization through the end of the RW Period
Long-Term Extension: Proportion of participants who maintained Clinical Response through the end of the LTE. | Up to 24 months
Long-Term Extension: Percentage of days with no or minimal pericarditis pain through the end of the LTE Period. | Up to 24 months
Long-Term Extension: Change from LTE Baseline in SF-36v2® Physical Component Summary score through the end of the LTE Period. | Up to 24 months
Long-Term Extension: Change from LTE Baseline in SF-36v2® Mental Component Summary score through the end of the LTE Period. | Up to 24 months
Long-Term Extension: Change from LTE baseline in pain NRS score through the end of the LTE Period. | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (30):
- United States (17):
  - Investigational Site 018, Gilbert, Arizona
  - Investigational Site 030, Los Angeles, California
  - Investigational Site 008, San Francisco, California
  - Investigational Site 016, Westminster, Colorado
  - Investigational Site 001, Columbus, Georgia
  - Investigational Site 004, Chicago, Illinois
  - Investigational Site 014, Indianapolis, Indiana
  - Investigational Site 002, Overland Park, Kansas
  - Investigational Site 012, Rochester, Minnesota
  - Investigational Site 015, New York, New York
  - Investigational Site 022, New York, New York
  - Investigational Site 009, Cincinnati, Ohio
  - Investigational Site 003, Cleveland, Ohio
  - Investigational Site 005, Austin, Texas
  - Investigational Site 013, Houston, Texas
  - Investigational Site 006, Charlottesville, Virginia
  - Investigational Site 023, Norfolk, Virginia
- Investigational Site 027, Ottawa, Ontario, Canada
- France (3):
  - Investigational Site 028, Montpellier
  - Investigational Site 021, Paris
  - Investigational Site 019, Poitiers
- Italy (2):
  - Investigational Site 029, Genoa
  - Investigational Site 007, Milan
- Serbia (2):
  - Investigational Site 025, Belgrade
  - Investigational Site 026, Belgrade
- Spain (3):
  - Investigational Site 010, Barcelona
  - Investigational Site 024, Madrid
  - Investigational Site 011, Murcia
- United Kingdom (2):
  - Investigational Site 020, London
  - Investigational Site 017, Southampton

IPD SHARING:
Plan to Share IPD: No